CLINICAL TRIAL: NCT03246126
Title: Visceral Manifold Study for the Repair of Thoracoabdominal Aortic Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-01441
Record Dates: First submitted 2017-08-02; First posted 2017-08-11 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: Thoracoabdominal Aortic Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Primary Arm: Treatment with Valiant Thoracoabdominal Stent Graft System (Experimental): The implantation of the Valiant Thoracoabdominal Stent Graft System is conducted under fluoroscopic/angiographic guidance.
  Interventions: Device: Valiant™Thoracoabdominal Stent Graft System
- Expanded Use Arm: Treatment with Valiant Thoracoabdominal Stent Graft System (Experimental): The implantation of the Valiant Thoracoabdominal Stent Graft System is conducted under fluoroscopic/angiographic guidance.
  Interventions: Device: Valiant™Thoracoabdominal Stent Graft System

INTERVENTIONS:
Device: Valiant™Thoracoabdominal Stent Graft System — The Visceral Manifold System is comprised of the Thoracic Bifurcation and Visceral Manifold to treat a thoracoabdominal aortic aneurysm or TAAA. The experimental procedure to implant the stent graft will be done in an operating room and will last anywhere from four to eight hours, but may take longer.
  Other Names: Endurant Stent Graft System

SUMMARY:
The purpose of this study is to evaluate the use of an investigational device called the ValiantTM Visceral Manifold Thoracoabdominal Stent Graft System for the repair of thoracoabdominal aortic aneurysms (TAAA), which is a balloon-like bulge in the aorta (major artery leading away from your heart) that originates in your chest and extends to your abdomen and also includes the branch arteries that supply blood to the liver, spleen, intestine, kidneys and other organs in your abdomen. The word "investigational" means the device is still being tested and is not approved by the Food and Drug Administration (FDA) for sale in the United States.

DETAILED DESCRIPTION:
The primary objective of the clinical investigation is to assess the use of the thoracic bifurcation and the visceral manifold to repair thoracoabdominal aortic aneurysms in patients having appropriate anatomy. The primary intent of the study is to assess safety (i.e. freedom from major adverse events (MAE) at 30 days) and preliminary effectiveness (i.e., treatment success and technical success) of the device (i.e., the proportion of treatment group subjects that achieve and maintain treatment success at one year). Additionally, the study will assess technical success and treatment success at each follow-up interval.

ELIGIBILITY:
Primary Arm Inclusion Criteria:

A patient may be entered into the study if the patient has at least one of the following

* An aneurysm with a maximum diameter of > 5.5 cm or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e., perpendicular to the centerline) measurements
* Aneurysm with a history of growth > 0.5 cm in 6 months
* Saccular aneurysm deemed at significant risk for rupture
* Symptomatic aneurysm greater than or equal to 4.5 cm

Additional Primary Arm Inclusion Criteria:

* Axillary or brachial and iliac or femoral access vessel morphology that is compatible with vascular access techniques, devices or accessories, with or without use of a surgical conduit
* Proximal landing zone for the thoracic bifurcation stent graft that has: (a) ≥ 2.5 cm of nonaneurysmal aortic segment including previously placed graft material (neck) distal to the left subclavian artery (LSA); (b) Diameter in the range of 26-42 mm; (c) Adequate distance from the celiac artery, in order to accommodate cannulation from the antegrade access point when considering the total deployed length of the thoracic bifurcation and visceral manifold
* Iliac artery or aortic distal fixation site, including both native tissue and previously placed graft, greater than or equal to 15 mm in length and diameter in the range of 8 - 25 mm
* Life expectancy: > 1 year

Expanded Use Arm Inclusion Criteria:

* Branch vessel diameter <5mm
* Urgent or emergent presentation
* Patient has a contained rupture
* Patient has a ruptured aneurysm
* Patient has a type B dissection (subacute or chronic) in the portion of the aorta intended to be treated
* Poor performance status including two major system failures (cardiovascular, pulmonary, renal, hepatobiliary, and neuromuscular)
* Baseline creatinine greater than 2.0 mg/dL
* Anatomy that does not allow maintenance of at least one hypogastric artery
* Anatomy that does not allow primary or assisted patency of the left subclavian artery
* Prior aneurysm repair that would involve relining of the previously placed graft material requiring placement of the investigational system in a landing zone that expands beyond any limits of the previously placed graft material
* Obstructive stenting of any or all of the visceral vessels
* Treatment of the patient population listed above will be considered for this expanded arm of the study if they are not a candidate for open surgical repair, cannot be treated with approved devices, and do not meet inclusion into the primary study arm as per opinion of the Principal Investigator, with the concurrence of the IRB.

Primary Arm Exclusion Criteria:

* Patient is a good candidate for and elects for open surgical repair
* Can be treated in accordance with the instructions for use with a legally marketed endovascular prosthesis
* Is eligible for enrollment in a manufacturer- sponsored IDE at the investigational site
* Unwilling to comply with the follow-up schedule
* Inability or refusal to give informed consent by patient or legal representative
* Urgent or emergent presentation
* Patient is pregnant or breastfeeding
* Patient has a contained rupture
* Patient has a ruptured aneurysm
* Patient has a dissection in the portion of the aorta intended to be treated
* Obstructive stenting of any or all of the visceral vessels
* Poor performance status including two major system failures (cardiovascular, pulmonary, renal, hepatobiliary, and neuromuscular)
* Prior aneurysm repair that would involve relining of the previously placed graft material requiring placement of the investigational system in a landing zone that expands beyond any limits of the previously placed graft material
* Known sensitivities or allergies to the materials of construction of the devices, including nitinol (Nickel: Titanium), polyester, platinum-iridium, polytetrafluoroethylene (PTFE), platinum, gold, polyethylene, or stainless steel.
* Known hypersensitivity or contraindication to anticoagulation or contrast media that cannot be adequately medically managed
* Uncorrectable coagulopathy
* Body habitus that would inhibit x-ray visualization of the aorta or exceeds the safe capacity of the equipment
* Patient has had a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned < 30 days of the endovascular repair
* Unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina)
* Systemic or local infection that may increase the risk of endovascular graft infection
* Baseline creatinine greater than 2.0 mg/dL
* History of connective tissue disorders (e.g., Marfan Syndrome, Ehler's Danlos Syndrome)
* ranch vessel diameter less than 5 mm
* Thrombus or excessive calcification within the neck of the aneurysm
* Anatomy that would not allow maintenance of at least one patent hypogastric artery
* Anatomy that would not allow primary or assisted patency of the left subclavian artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Maldonado, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 individuals were enrolled in the study; however, 7 of these individuals did not start the study. Thus, the total number of participants who started the study is n=10.
Period: Overall Study
Arm/Group | Primary Arm: Treatment With Valiant Thoracoabdominal Stent Graft System | Expanded Use Arm: Treatment With Valiant Thoracoabdominal Stent Graft System
Started | 5 | 5
Completed | 5 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Arm: Treatment With Valiant Thoracoabdominal Stent Graft System | Expanded Use Arm: Treatment With Valiant Thoracoabdominal Stent Graft System | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (7) | 67.6 (15.6) | 70.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Major Adverse Events (MAE) at Day 30
Description: Freedom from MAE is defined as the number of participants who have not experienced a major adverse event (including death, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, and stroke) at 30 days.
Time Frame: Up to Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Arm: Treatment With Valiant Thoracoabdominal Stent Graft System | Expanded Use Arm: Treatment With Valiant Thoracoabdominal Stent Graft System
Number analyzed (Participants) | 5 | 5
Participants | 3 | 4

2. Primary Outcome: Number of Participants Who Achieve Technical Success
Description: Technical success is defined as successful access of the aneurysm site and deployment of the Visceral Manifold investigational devices in intended locations.
Time Frame: Up to Year 1
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Arm: Treatment With Valiant Thoracoabdominal Stent Graft System | Expanded Use Arm: Treatment With Valiant Thoracoabdominal Stent Graft System
Number analyzed (Participants) | 5 | 4
Participants | 5 | 4

3. Secondary Outcome: Freedom From Paraplegia at Day 30
Description: Number of participants who have not experienced paraplegia at Day 30.
Time Frame: Up to Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Arm: Treatment With Valiant Thoracoabdominal Stent Graft System | Expanded Use Arm: Treatment With Valiant Thoracoabdominal Stent Graft System
Number analyzed (Participants) | 5 | 5
Participants | 3 | 4

ADVERSE EVENTS:
Time Frame: 5 years
Description: Assessed via physical examination, blood samples, metabolic panel, and other tests at follow-up visits.
Arm/Group | Primary Arm: Treatment With Valiant Thoracoabdominal Stent Graft System | Expanded Use Arm: Treatment With Valiant Thoracoabdominal Stent Graft System
All-Cause Mortality (participants affected / at risk) | 4/5 | 3/5
Serious Adverse Events (participants affected / at risk) | 5/5 | 4/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Arm: Treatment With Valiant Thoracoabdominal Stent Graft System (N=5) | Expanded Use Arm: Treatment With Valiant Thoracoabdominal Stent Graft System (N=5)
Paraplegia (Musculoskeletal and connective tissue disorders) | 2 | 1
Renal Failure (Renal and urinary disorders) | 0 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Acute Cholecystitis (Hepatobiliary disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Celiac Occlusion (Gastrointestinal disorders) | 1 | 0
Clot (Mural Thrombus) (Vascular disorders) | 0 | 1
Congestive Heart Failure (Cardiac disorders) | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0
Endoleak Type 1b (Injury, poisoning and procedural complications) | 2 | 1
Endoleak Type 1c Left Renal Stent (Injury, poisoning and procedural complications) | 0 | 1
Endoleak Type 3 Left Renal (Injury, poisoning and procedural complications) | 0 | 1
Endoleak Type Iii (Injury, poisoning and procedural complications) | 0 | 1
Enlarging Aneurysmal Sac (Injury, poisoning and procedural complications) | 0 | 1
Exacerbation Of Respiratory Distress Due To Covid (Infections and infestations) | 1 | 0
Extremities - Arterial Insufficiency Or Ischemia (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Left Femoral Artery Access Injury (Injury, poisoning and procedural complications) | 0 | 1
Loss Of Seal Of Left Common Iliac Artery (Cia) (Injury, poisoning and procedural complications) | 1 | 0
Methicillin-Sensitive Staphylococcus Aureus (Infections and infestations) | 1 | 0
Multi Organ Failure (General disorders) | 0 | 1
Neurogenic Bladder (Nervous system disorders) | 2 | 0
Neurogenic Bowel (Nervous system disorders) | 2 | 0
Paraparesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumoperitoneum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumoperitoneum Ii (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Vascular disorders) | 0 | 1
Right Renal Stent Occlusion (Injury, poisoning and procedural complications) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic Shock With Bacteremia (Infections and infestations) | 0 | 1
Significant Intra-Operative Bleeding (Injury, poisoning and procedural complications) | 0 | 1
Staphlococcus Aureus Bacteremia Secondary To Sacral Ulcer (Infections and infestations) | 0 | 1
Superior Mesenteric Artery Occlusion (Vascular disorders) | 1 | 0
Upper GI Bleed (Gastrointestinal disorders) | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Arm: Treatment With Valiant Thoracoabdominal Stent Graft System (N=5) | Expanded Use Arm: Treatment With Valiant Thoracoabdominal Stent Graft System (N=5)
1st Degree Atrioventricular (AV) Block (Cardiac disorders) | 1 | 0
Abscess Under Sacral Ulcer (Infections and infestations) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 0
Acute Subarachnoid Hemorrhage (Vascular disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 4 | 4
Anemia (Post Op) (Blood and lymphatic system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Atelectasis-Left (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Bell's Palsy (Nervous system disorders) | 0 | 1
Bilateral Groin Hematomas (Vascular disorders) | 1 | 0
Bilateral Hip Wounds (Injury, poisoning and procedural complications) | 1 | 0
Bilateral Hydronephrosis (Renal and urinary disorders) | 0 | 1
Bilateral Inguinal Hematoma (Vascular disorders) | 0 | 1
Bilateral Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Bilateral Subdural Hematoma (Vascular disorders) | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Chronic Constipation (Gastrointestinal disorders) | 1 | 0
Chronic Renal Failure (Renal and urinary disorders) | 0 | 1
Cyst Left Kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Decubitus Ulcer (General disorders) | 0 | 1
Demand Ischemia/Elevated Troponin (Cardiac disorders) | 1 | 0
Dissection Of Left Axillary Artery (Surgical and medical procedures) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Deep vein thrombosis (DVT) (Vascular disorders) | 0 | 1
Edema Posterior Paraspinal Musculature (General disorders) | 1 | 0
Edema-Lower Extremities (General disorders) | 1 | 0
Endoleak Stable Type 2 (Injury, poisoning and procedural complications) | 0 | 1
Endoleak Type 2 (Injury, poisoning and procedural complications) | 1 | 1
Endoleak Type 2 (Stable) (Injury, poisoning and procedural complications) | 1 | 0
Fever (General disorders) | 0 | 2
Gallbladder Distention (Gastrointestinal disorders) | 1 | 0
Gluteal Hematoma (Vascular disorders) | 1 | 0
Gluteal Wound (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hearing Loss (Ear and labyrinth disorders) | 0 | 1
Hematoma Spinal Drain Site (Vascular disorders) | 0 | 1
Hematoma X 2 Left Upper Arm (Vascular disorders) | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hepatic Artery Extravasation Dissection (Surgical and medical procedures) | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Hypervolemia (Blood and lymphatic system disorders) | 0 | 1
Hyponatremia (Blood and lymphatic system disorders) | 1 | 1
Intermittent Atrial Fibrillation (Cardiac disorders) | 0 | 1
Intermittent Confusion (Psychiatric disorders) | 1 | 0
Intermittent Urinary Retention (Renal and urinary disorders) | 1 | 0
Intraoperative Blood Loss (Injury, poisoning and procedural complications) | 0 | 1
Left Atrial Dilatation (Cardiac disorders) | 0 | 1
Left Axillary Fluid Collection (General disorders) | 1 | 0
Left Lobe Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Moderate-Severe Mid Right Coronary Artery Disease (Cardiac disorders) | 0 | 1
Neurogenic Bladder (Nervous system disorders) | 0 | 1
Neurogenic Bowel (Nervous system disorders) | 0 | 1
Neurogenic Ileus (Nervous system disorders) | 0 | 1
Penile Edema (Reproductive system and breast disorders) | 1 | 0
Penile Ulcer (Reproductive system and breast disorders) | 1 | 0
Penile/Scrotal Edema (Reproductive system and breast disorders) | 0 | 1
Pleural Effusion Left (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postoperative Anemia (Blood and lymphatic system disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Progression Of Metastatic Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pulmonary Hypertension (Vascular disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash-Lace Pattern-Feet (Skin and subcutaneous tissue disorders) | 1 | 0
Renal Stone (Renal and urinary disorders) | 1 | 0
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Right Heel Ulcer (General disorders) | 1 | 0
Right Heel Wound (Injury, poisoning and procedural complications) | 1 | 0
Sacral Wound (Injury, poisoning and procedural complications) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus Bradycaria (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Situational Depression (Psychiatric disorders) | 1 | 0
Small Splenic Infarct (Vascular disorders) | 1 | 0
Splenic Infarct (Vascular disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 3
Toxic Metabolic Encephalopathy (Metabolism and nutrition disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT03246126/Prot_SAP_000.pdf